CLINICAL TRIAL: NCT02354326
Title: Evaluation of Bone Metastases With Dual Energy Computed Tomography (CT)
Brief Title: Dual Energy Computed Tomography (CT) in Finding Bone Metastases in Patients With Cancer
Status: Terminated | Type: Observational
Why Stopped: No bone lesions detected and poor accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE5Y14; NCI-2014-02497 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE5Y14 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-01-28; First posted 2015-02-03 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Malignant Neoplasm; Metastatic Malignant Neoplasm to the Bone
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic (VNC DECT): Patients undergo CT scans. Additional images will be processed with virtual non-calcium (VNC) dual energy CT (DECT) information. Comparison will be made between images with and without addition of VNC.
  Interventions: Radiation: virtual non-calcium dual-energy computed tomography; Radiation: computed tomography

INTERVENTIONS:
Radiation: virtual non-calcium dual-energy computed tomography — Undergo VNC DECT
  Other Names: VNC DECT
Radiation: computed tomography — Undergo CT without VNC
  Other Names: CT

SUMMARY:
This clinical trial studies dual energy computed tomography (CT) in finding cancer that has spread from the original (primary) tumor to the bone (bone metastases) in patients with cancer. Diagnostic procedures, such as dual energy CT, may help find and diagnose bone metastases and may be more accurate compared to single energy CT alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the accuracy of single energy CT (SECT) with virtual non-calcium (VNC) double energy CT (DECT) to standard SECT alone in the detection of metastatic bone lesions using positron emission tomography (PET)-CT as the reference standard.

OUTLINE:

Computed tomography (CT) scans are routinely used in the evaluation of oncologic patients for initial diagnosis and subsequent disease staging. Detection of bone metastasis on standard CT, however, is limited in sensitivity, particularly in case of osteolytic intramedullary lesions. Recent studies have shown the ability to detect bone marrow edema using CT with the use of a virtual non-calcium (VNC) dual energy CT (DECT) technique. Because bone marrow edema is similar in composition to intramedullary bone metastases (i.e. both are of soft tissue composition as opposed to calcium or fat), VNC DECT may also be helpful in the detection of bone marrow metastasis. Cancer patients obtaining a Positron Emission Tomography (PET) CT and a separate diagnostic CT scan as part of their routine clinical care will be enrolled into the study. The diagnostic CT scan will be performed on a DECT scanner and the images will be reconstructed as SECT images for routine clinical interpretation as well as VNC DECT images. The SECT images alone will be evaluated and scored, and then the VNC DECT images will be added to the SECT images for a second evaluation (consecutive reading session). Multiple readers blinded to the PET-CT findings for detection of bony metastatic disease will participate.

Researchers hypothesize the addition of VNC DECT to SECT will be more accurate in the detection of metastatic bone marrow lesions compared to SECT alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients being imaged with PET/CT for diagnosis and/or staging of disease at Case Comprehensive Cancer Center
* Patients with bone metastases on PET/CT
* Patients without bone metastases on PET/CT
* All cancer types and both newly diagnosed and previously treated patients will be included

Exclusion Criteria:

* Patients with intervening treatment during the time between diagnostic CT and PET/CT
* Time between the diagnostic CT and PET/CT greater than 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients obtaining a Positron Emission Tomography (PET) CT and a separate diagnostic CT scan as part of their routine clinical care
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2017-09-27 (Actual); Study Completion 2017-09-27 (Actual)

PRIMARY OUTCOMES:
Number of Lesions Present | within 30 days of first treatment
  Number of lesions detected at the 46 designated locations at the time of the VNC DECT
Number of lesions absent | within 30 days of first treatment
  Number of absent lesions from the 46 designated locations at the time of the VNC DECT
Confidence in the presence of one or more lesions in that particular anatomic location using a 0-100 point confidence scale | within 30 days of first treatment
  Each location will be correlated with PETCT which will serve as the reference standard.
Accuracy of VNC DECT | within 30 days of first treatment
  Will be measured using nonparametric estimates of the area under the receiver operating characteristic (ROC) curve using methods for clustered data (i.e. multiple locations per patient). ROC area estimates will be constructed for each reader for both SECT alone and DECT as an adjunct to SECT. For each reader, the ROC areas of SECT and DECT plus SECT will be compared using a Wald test; a significance level of 0.05 will be used. Analysis of variance methods for multiple-reader ROC studies will be used. A 95% confidence interval for the difference in ROC areas will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Subhas, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02354326/Prot_SAP_000.pdf